CLINICAL TRIAL: NCT06785051
Title: Effects of AI-Based Physiotherapy on Mandibular Mobility, Shoulder Function, Whole-Body Physical Function, and Quality of Life in Oral Cancer Patients
Brief Title: AI-based Physiotherapy for Oral Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202411044RINC
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-12

CONDITIONS: Oral Cancer
Keywords: Artificial intelligence; Oral cancer; Maximum interincisal opening; Physical function; Prehabilitation; Physiotherapy
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): AI-based physiotherapy
  Interventions: Behavioral: AI-based physiotherapy; Behavioral: Scar management
- Control group (Active Comparator): Usual care
  Interventions: Behavioral: Conventional physiotherapy; Behavioral: Scar management

INTERVENTIONS:
Behavioral: AI-based physiotherapy — jaw, neck, shoulder ROM exercises, and scapular-focused exercises guided by AI technology, 30 minutes of intervention, once a week, and a total of 12 weeks
  Arms: Experimental group
Behavioral: Conventional physiotherapy — jaw, neck, shoulder ROM exercises, and scapular-focused exercises, 30 minutes of intervention, once a week, and a total of 12 weeks
  Arms: Control group
Behavioral: Scar management — scar massage and jaw-mobilizing exercises combined with devices or depressors

SUMMARY:
This study examines the effects of AI-based physiotherapy on oral function, shoulder function, whole-body physical function, and quality of life in oral cancer patients. One hundred patients will be recruited before surgery, chemotherapy, or radiotherapy and randomly assigned to an experimental group receiving 12 weeks of AI-guided physiotherapy or a control group receiving usual care. Both groups will perform jaw, neck, and shoulder exercises, with the experimental group using a mobile app to monitor progress. Assessments at baseline, pre-intervention, and 3 months post-intervention will measure maximal in the maximum interincisal opening (MIO), joint range of motion (ROM), pain, endurance (e.g., 6-minute walk test), upper extremity function, and quality of life.

DETAILED DESCRIPTION:
This study examines the effects of AI-based physiotherapy on oral function (e.g., mouth opening), shoulder function (e.g., shoulder joint range of motion and upper extremity function), whole-body physical function (e.g., 6-minute walk test), and health-related quality of life. 100 newly diagnosed oral cancer patients will be recruited before surgery, chemotherapy, or radiotherapy and randomly assigned to two groups. The experimental group will receive AI-based physiotherapy for 12 weeks, including postural correction exercises guided by AI technology, while the control group will receive usual care. Both groups will perform jaw, neck, and shoulder exercises, with the experimental group using a mobile app to monitor progress and record their exercise diaries. Assessments at baseline, pre-intervention, and 3 months post-intervention will measure the maximum interincisal opening (MIO), joint range of motion (ROM), pain, endurance, and upper extremity function using the Disabilities of the Arm, Shoulder, and Hand (DASH) scores, and quality of life using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed oral cancer patients who are scheduled to receive cancer-related treatments (e.g., oral cancer surgery, radiotherapy, chemotherapy, or chemoradiotherapy).
* Age between 20 and 65 years.

Exclusion Criteria:

* Could not communicate.
* Had any disorder that could influence movement performance.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in maximal mouth opening | baseline, pre-intervention, 3-months post-intervention
  Average maximal mouth opening measured 3 times in mm
Change from baseline in shoulder joint range of motion | baseline, pre-intervention, 3-months post-intervention
  Average range of motion of shoulder abduction measured 3 times in degrees

SECONDARY OUTCOMES:
Change from baseline in function on Disabilities of the Arm, Shoulder, and Hand outcome questionnaire | baseline, pre-intervention, 3-months post-intervention
  A total scale from 1 to 100. Higher scores indicate greater disability.
Change from baseline in health-related function on EORTC QLQ-C30 questionnaire | baseline, pre-intervention, 3-months post-intervention
  A total scale from 1 to 100. Higher scores indicate greater function.
Change from baseline in whole-body physical function on 6-minute walk test | baseline, pre-intervention, 3-months post-intervention
  Walking distance measured in meters.
Change from baseline in shoulder pain | baseline, pre-intervention, 3-months post-intervention
  Visual analog scale from 0 to 10. Higher scores indicate most pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — National Taiwan University, College of Medicine
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Background] Loos H, Sahm H, Sprenger GA. Glucose-fructose oxidoreductase, a periplasmic enzyme of Zymomonas mobilis, is active in its precursor form. FEMS Microbiol Lett. 1993 Mar 1;107(2-3):293-8. doi: 10.1111/j.1574-6968.1993.tb06045.x. PMID 8472911
- [Background] Baranano CF, Rosenthal EL, Morgan BA, McColloch NL, Magnuson JS. Dynasplint for the management of trismus after treatment of upper aerodigestive tract cancer: a retrospective study. Ear Nose Throat J. 2011 Dec;90(12):584-90. doi: 10.1177/014556131109001209. PMID 22180114
- [Background] Chen CC, Lin CC, Hsieh HP, Fu YC, Chen YJ, Lu TW. In vivo three-dimensional mandibular kinematics and functional point trajectories during temporomandibular activities using 3d fluoroscopy. Dentomaxillofac Radiol. 2021 Feb 1;50(2):20190464. doi: 10.1259/dmfr.20190464. Epub 2020 Aug 12. PMID 32783637
- [Background] Chen SC, Huang BS, Hung TM, Lin CY, Chang YL. Impact of physical and psychosocial dysfunction on return to work in survivors of oral cavity cancer. Psychooncology. 2019 Sep;28(9):1910-1917. doi: 10.1002/pon.5173. Epub 2019 Jul 23. PMID 31291694
- [Background] Chen YH, Liang WA, Lin CR, Huang CY. A randomized controlled trial of scapular exercises with electromyography biofeedback in oral cancer patients with accessory nerve dysfunction. Support Care Cancer. 2022 Oct;30(10):8241-8250. doi: 10.1007/s00520-022-07263-4. Epub 2022 Jul 11. PMID 35821447
- [Background] Chen YH, Huang CY, Liang WA, Lin CR, Chao YH. Effects of Conscious Control of Scapular Orientation in Oral Cancer Survivors With Scapular Dyskinesis: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211040827. doi: 10.1177/15347354211040827. PMID 34412536
- [Background] Chen YH, Lin CR, Liang WA, Huang CY. Motor control integrated into muscle strengthening exercises has more effects on scapular muscle activities and joint range of motion before initiation of radiotherapy in oral cancer survivors with neck dissection: A randomized controlled trial. PLoS One. 2020 Aug 6;15(8):e0237133. doi: 10.1371/journal.pone.0237133. eCollection 2020. PMID 32760097
- [Background] Chen YH, Liang WA, Hsu CY, Guo SL, Lien SH, Tseng HJ, Chao YH. Functional outcomes and quality of life after a 6-month early intervention program for oral cancer survivors: a single-arm clinical trial. PeerJ. 2018 Feb 21;6:e4419. doi: 10.7717/peerj.4419. eCollection 2018. PMID 29492348
- [Background] Cocks K, Wells JR, Johnson C, Schmidt H, Koller M, Oerlemans S, Velikova G, Pinto M, Tomaszewski KA, Aaronson NK, Exall E, Finbow C, Fitzsimmons D, Grant L, Groenvold M, Tolley C, Wheelwright S, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group. Content validity of the EORTC quality of life questionnaire QLQ-C30 for use in cancer. Eur J Cancer. 2023 Jan;178:128-138. doi: 10.1016/j.ejca.2022.10.026. Epub 2022 Nov 1. PMID 36436330
- [Background] Cohen EE, LaMonte SJ, Erb NL, Beckman KL, Sadeghi N, Hutcheson KA, Stubblefield MD, Abbott DM, Fisher PS, Stein KD, Lyman GH, Pratt-Chapman ML. American Cancer Society Head and Neck Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 May;66(3):203-39. doi: 10.3322/caac.21343. Epub 2016 Mar 22. PMID 27002678
- [Background] Dijkstra PU, Huisman PM, Roodenburg JL. Criteria for trismus in head and neck oncology. Int J Oral Maxillofac Surg. 2006 Apr;35(4):337-42. doi: 10.1016/j.ijom.2005.08.001. Epub 2005 Nov 8. PMID 16280237
- [Background] Falz R, Bischoff C, Thieme R, Lassing J, Mehdorn M, Stelzner S, Busse M, Gockel I. Effects and duration of exercise-based prehabilitation in surgical therapy of colon and rectal cancer: a systematic review and meta-analysis. J Cancer Res Clin Oncol. 2022 Sep;148(9):2187-2213. doi: 10.1007/s00432-022-04088-w. Epub 2022 Jun 13. PMID 35695931
- [Background] Furtado DA, Pereira AA, Andrade Ade O, Bellomo DP Jr, da Silva MR. A specialized motion capture system for real-time analysis of mandibular movements using infrared cameras. Biomed Eng Online. 2013 Feb 22;12:17. doi: 10.1186/1475-925X-12-17. PMID 23433470
- [Background] Jehn P, Spalthoff S, Lentge F, Zeller AN, Tavassol F, Neuhaus MT, Eckstein FM, Kruskemper G, Gellrich NC, Korn P. Postoperative quality of life and therapy-related impairments of oral cancer in relation to time-distance since treatment. J Cancer Surviv. 2022 Dec;16(6):1366-1378. doi: 10.1007/s11764-021-01118-3. Epub 2021 Oct 5. PMID 34609700
- [Background] Johnson J, Johansson M, Ryden A, Houltz E, Finizia C. Impact of trismus on health-related quality of life and mental health. Head Neck. 2015 Nov;37(11):1672-9. doi: 10.1002/hed.23816. Epub 2015 Jan 27. PMID 24985733
- [Background] Kamstra JI, Reintsema H, Roodenburg JL, Dijkstra PU. Dynasplint Trismus System exercises for trismus secondary to head and neck cancer: a prospective explorative study. Support Care Cancer. 2016 Aug;24(8):3315-23. doi: 10.1007/s00520-016-3131-4. Epub 2016 Mar 8. PMID 26956713
- [Background] Li YH, Chang WC, Chiang TE, Lin CS, Chen YW. Mouth-opening device as a treatment modality in trismus patients with head and neck cancer and oral submucous fibrosis: a prospective study. Clin Oral Investig. 2019 Jan;23(1):469-476. doi: 10.1007/s00784-018-2456-4. Epub 2018 Apr 26. PMID 29696422
- [Background] Loewen I, Jeffery CC, Rieger J, Constantinescu G. Prehabilitation in head and neck cancer patients: a literature review. J Otolaryngol Head Neck Surg. 2021 Jan 6;50(1):2. doi: 10.1186/s40463-020-00486-7. PMID 33407922
- [Background] Marinelli F, Lezcano MF, Alarcon J, Navarro P, Fuentes R. A Novel Technique to Accurately Measure Mouth Opening Using 3D Electromagnetic Articulography. Bioengineering (Basel). 2022 Oct 19;9(10):577. doi: 10.3390/bioengineering9100577. PMID 36290545
- [Background] McMillan H, Barbon CEA, Cardoso R, Sedory A, Buoy S, Porsche C, Savage K, Mayo L, Hutcheson KA. Manual Therapy for Patients With Radiation-Associated Trismus After Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):418-425. doi: 10.1001/jamaoto.2022.0082. PMID 35297966
- [Background] Michael CM, Lehrer EJ, Schmitz KH, Zaorsky NG. Prehabilitation exercise therapy for cancer: A systematic review and meta-analysis. Cancer Med. 2021 Jul;10(13):4195-4205. doi: 10.1002/cam4.4021. Epub 2021 Jun 10. PMID 34110101
- [Background] Pauli N, Svensson U, Karlsson T, Finizia C. Exercise intervention for the treatment of trismus in head and neck cancer - a prospective two-year follow-up study. Acta Oncol. 2016 Jun;55(6):686-92. doi: 10.3109/0284186X.2015.1133928. Epub 2016 Feb 15. PMID 26878553
- [Background] Shao CH, Chiang CC, Huang TW. Exercise therapy for cancer treatment-induced trismus in patients with head and neck cancer: A systematic review and meta-analysis of randomized controlled trials. Radiother Oncol. 2020 Oct;151:249-255. doi: 10.1016/j.radonc.2020.08.024. Epub 2020 Sep 3. PMID 32890607
- [Background] van der Geer SJ, Reintsema H, Kamstra JI, Roodenburg JLN, Dijkstra PU. The use of stretching devices for treatment of trismus in head and neck cancer patients: a randomized controlled trial. Support Care Cancer. 2020 Jan;28(1):9-11. doi: 10.1007/s00520-019-05075-7. Epub 2019 Nov 7. PMID 31701267
- [Background] Watters AL, Cope S, Keller MN, Padilla M, Enciso R. Prevalence of trismus in patients with head and neck cancer: A systematic review with meta-analysis. Head Neck. 2019 Sep;41(9):3408-3421. doi: 10.1002/hed.25836. Epub 2019 Jun 19. PMID 31215723